CLINICAL TRIAL: NCT05131035
Title: Targeting Processing Speed Deficits to Improve Social Functioning and Lower Psychosis Risk in Adolescents at Clinical High Risk for Psychosis
Brief Title: Targeting Processing Speed Deficits to Improve Social Functioning and Lower Psychosis Risk
Acronym: SCORES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 21-0832, 23-0500; R61MH123574 (NIH); R33MH123574 (NIH)
Record Dates: First submitted 2021-11-11; First posted 2021-11-23 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Psychosis; Prodromal Schizophrenia; Prodromal Symptoms
Keywords: Clinical High Risk (CHR); Processing Speed; Social Functioning; Social Impairment; Social Skills; Adolescents; Cognitive Remediation
MeSH Terms: conditions — Psychotic Disorders; Schizotypal Personality Disorder; Prodromal Symptoms; Social Adjustment; Social Skills | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: The R33 study design will utilize a randomized intervention model. All participants will participate in cognitive training with small group support.One group will complete speeded cognitive training tasks and the other group will complete non-speeded cognitive training tasks.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Speeded Cognitive Training (Experimental): Participants in this condition will complete 40 hours of Cognitive Remediation with a mid-point assessment (20 hours/5 weeks) to determine the impact of speeded cognitive training tasks on cognition and social function.
  Interventions: Behavioral: SCORES (Specific COgnitive Remediation with Support)
- Non-Speeded Cognitive Training (Active Comparator): Participants in this condition will complete 40 hours of Cognitive Remediation with a mid-point assessment (20 hours/5 weeks) to determine the impact of non-speeded cognitive training tasks on cognition and social function.
  Interventions: Behavioral: SCORES (Specific COgnitive Remediation with Support)

INTERVENTIONS:
Behavioral: SCORES (Specific COgnitive Remediation with Support) — This study evaluates the effectiveness of a 10-week cognitive remediation program plus group coaching and therapy to improve processing speed and, in turn, social functioning and attenuated positive symptoms in CHR subjects. The SCORES (Specific COgnitive Remediation with Support) intervention is a novel CR program combined with group coaching, performance-based rewards, game-like tasks, and therapy elements to increase engagement and retention.
  In the 2 year, R61 phase, all participants will complete 40 hours of CR (4 hrs per week) with a mid-point assessment (20 hours of CR at 5 weeks) to determine the impact of CR on processing speed as measured by the MCCB.
  The second phase of the study (R33) will compare the 40 hours of speeded brain training to 40 hours of non-speeded brain training. This three year study will allow for a replication and assessment of specificity of the targeted intervention.

SUMMARY:
This 10 week intervention, Specific Cognitive Remediation with Surround (or SCORES), is designed to target processing speed, a cognitive domain related directly to social functioning, which in turn, represents a vulnerability factor for psychosis. This remotely-delivered intervention combining targeted cognitive training exercises and group support was developed to directly impact processing speed, and at the same time, boost motivation and engagement in adolescents at risk for schizophrenia and other psychotic disorders.

DETAILED DESCRIPTION:
This study evaluates the effectiveness of a cognitive remediation (CR) program plus group coaching and support designed to improve processing speed and, in turn, social functioning and attenuated positive symptoms in individual considered Clinical High Risk for psychosis. The SCORES (Specific COgnitive REmediation with Support) intervention is a novel Cognitive Remediation program combined with group coaching, performance-based rewards, game-like tasks, and educational elements to increase engagement and retention. The study is funded by a R61/R33 award. In the R61 phase, all participants were asked to complete 40 hours of Cognitive Remediation or brain training (4 hours per week/10 weeks) with a mid-point assessment (at 5 weeks) to determine the training dose needed to impact processing speed as measured by the Matrics Cognitive Consensus Battery. The current R33 (Phase 2) will look to replicate the results of the R61 and assess the specificity of the targeted intervention with the addition of a non-speeded cognitive training group..

ELIGIBILITY:
Inclusion Criteria:

* Meet Clinical High Risk (CHR) criteria on the Structured Interview for Psychosis Risk Syndromes, defined by the presence of at least one attenuated positive symptom at a moderate to severe level
* A score representing 0.5 SD below the mean on Animal Naming, Trails A or BACS: Symbol Coding from the MATRICS Consensus Cognitive Battery (MCCB).

Exclusion Criteria:

* Any DSM 5 Schizophrenia-Spectrum diagnosis
* Non-English speaking
* Past or current history of a clinically significant central nervous system disorder (e.g., seizure disorder)
* Estimated IQ<70
* Significant head injury
* Significant substance abuse
* Significant visual or auditory impairment.

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-10-28 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Processing Speed domain score from the MATRICS Consensus Cognitive Battery (MCCB) | Baseline, Mid-Treatment (5 weeks), Post Treatment (10 weeks)
  Change in processing speed domain score and individual measures within the domain.

SECONDARY OUTCOMES:
Global Functioning: Social (GF:Social) scale (Phase 2/R33 only) | Baseline, Mid-Treatment (5 weeks), Post Treatment (10 weeks)
  Change in GF:Social score from baseline to follow up timepoints. The GF:Social scale scores range from 1 to 10 with higher scores representing better social functioning.
SIPS/SOPS: Positive Symptoms (Phase 2/R33 only) | Baseline, Mid-Treatment (5 weeks), Post Treatment (10 weeks)
  Change in Total Positive Symptom score from baseline to follow up timepoints. Each of the 5 positive symptoms on the SOPS range from 0-6 (6 indicating a psychotic symptom).

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo E Carrion, Ph.D., Principal Investigator — Northwell Health
Locations (1):
- Northwell Health- The Zucker Hillside Hospital, Glen Oaks, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be uploaded to the NIH Data Archive (NDA).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: We plan to make all data collected available as a national resource to the broader scientific community for investigators wishing to pursue their own analyses. Consistent with the NIH policy regarding data sharing, we will share data no later than following acceptance for publication of the main findings from the final dataset, which is expected to occur at the end of year 5. We request that we maintain exclusive access to these data until the end of year 5 to ensure an adequate amount of time for the PIs to conduct analyses and prepare manuscripts for publication. All de-identified data resulting from this NIH-funded award will be submitted to the NIMH Data Archive (NDA) according to this timeline, along with appropriate supporting documentation to enable efficient use of the data by other researchers not involved in the study. Data derived from the proposed study will also be shared through presentation at research conferences and through publication in peer-reviewed journals.
Access Criteria: Data will be shared with researchers upon request. Other researchers across the world can then request the pseudo-anonymized study data for other research from the NDA. Every researcher (and institutions to which they belong) who requests the pseudo-anonymized study data must promise to keep the data safe. Experts at the NIH will review each request carefully to reduce risks to participant privacy.